CLINICAL TRIAL: NCT04347928
Title: Respiratory and Hemodynamic Changes Induced in Mechanically Ventilated Patients for COVID-19
Acronym: PHYSIO-COVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_32; 2020-A00957-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; ARDS; Sars-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the present context, it seems necessary to try to describe as precisely as possible the physiological alterations due to COVID-19. From these observations, therapeutic proposals adapted to this new disease may then be developed, particularly in the symptomatic management of the critically ill patient. It therefore seems essential to rigorously study these modifications, as they have been studied in the past for ARDS.

The aim of this non-interventional study is to describe precisely the respiratory and hemodynamic changes induced by COVID-19 in mechanically ventilated patients

.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in intensive care for a SARS-CoV2 infection
* requiring invasive ventilation,
* intubated for less than 72 hours with PaO2/FiO2 ratio < 200 mmHg

Exclusion Criteria:

* Patient mechanically ventilated for 72 hours or more
* Patient with documented respiratory co-infection
* Patient with a contraindication to pulmonary artery catheter insertion: High risk of bleeding, pre-existing high degree of atrioventricular heart block , Pace Maker
* Patient with spontaneous ventilation
* Patient with severe ARDS with static compliance of the respiratory system < 20 mL/cmH2O
* Patient with severe ARDS with indication of prone positioning at inclusion.
* Patient with a cardiac condition that renders the measurement of pulmonary artery occlusion pressure uninterpretable as a surrogate for left ventricle end diastolic pressure (severe mitral insufficiency, severe mitral stricture, severe aortic insufficiency).
* Patient with intracardiac shunt
* Patient with ECMO
* Minors and pregnant women.
* Person not affiliated to or not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient hospitalized in ICU mechanically ventilated for less than 72 hours
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
intrapulmonary shunt ratio | during ICU stay, in the first 72 hours of mechanical ventilation initiation

SECONDARY OUTCOMES:
Evolution of respiratory variables | during ICU stay, in the first 72 hours of mechanical ventilation initiation
  Evaluation of PaO2 variation between in a high level of PEEP (15cmH2O) and a low level of PEEP (5cmH2O)
Evolution of respiratory variables | during ICU stay, in the first 72 hours of mechanical ventilation initiation
  Evaluation of PaCO2 variation between in a high level of PEEP (15cmH2O) and a low level of PEEP (5cmH2O)
Evolution of hemodynamic stability variables | during ICU stay, in the first 72 hours of mechanical ventilation initiation
  Evaluation of cardiac output variation between a high level of PEEP (15cmH2O) and a low level of PEEP (5cmH2O)

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Duburcq, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France